CLINICAL TRIAL: NCT04611204
Title: Prevalence of Transthyretin Cardiac Amyloidosis in Patients With Idiopathic Carpal Tunnel Syndrome Referred for Release Surgery
Brief Title: Transthyretin Cardiac Amyloidosis in Patients With Idiopathic Carpal Tunnel Syndrome Referred for Release Surgery
Acronym: PRATHYC
Status: Terminated | Type: Observational
Why Stopped: insufficient recruitment
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/18/0470
Record Dates: First submitted 2020-10-26; First posted 2020-11-02 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Transthyretin Amyloidosis; Carpal Tunnel Syndrome
Keywords: cardiac amyloidosis; transthyretin amyloidosis; carpal tunnel syndrome
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related; Carpal Tunnel Syndrome; Amyloid Neuropathies, Familial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Descriptive cohort — NT-proBNP assay, electrocardiogram and transthoracic echocardiography before CTS surgery release. Pathological analysis for amyloid deposits of transverse carpal ligament of patients included.

SUMMARY:
This study will determine the prevalence of transthyretin amyloidosis in pathology of the transverse carpal ligament and cardiac involvement using natriuretic peptides, electrocardiography and echocardiography in patients referred for carpal tunnel release surgery of idiopathic carpal tunnel syndrome. This study will describe the relationship between amyloid deposition observed on the transverse carpal ligament and the presence of cardiac involvement.

DETAILED DESCRIPTION:
Unrecognized wild-type transthyretin amyloidosis (ATTRwt) in patients with idiopathic carpal tunnel syndrome (CTS) is a prevalent aging-related disorder. Amyloid deposition in the tenosynovial tissue has been reported in ~35% of patients with idiopathic carpal tunnel syndrome.

Otherwise, CTS has been shown to be the most common initial symptom of systemic wild-type transthyretin amyloidosis. The clinical significance of subclinical ATTRwt deposits in the heart in elderly patients has yet to be determined, but these deposits could contribute to the development of heart failure with preserved ejection fraction. ATTRwt has been reported in ~15% of patients with heart failure with preserved ejection fraction. Early detection of amyloid deposition in the transverse carpal ligament of patients with CTS could anticipate cardiac damage and progression to heart failure.The aim of this study is to determine the prevalence of transthyretin amyloidosis in pathology of the transverse carpal ligament and cardiac involvement using natriuretic peptides, electrocardiography and echocardiography in patients referred for carpal tunnel release surgery of idiopathic carpal tunnel syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 year-old
* Indication carpal tunnel release surgery of idiopathic carpal tunnel syndrome.
* To agree to participate (signature of the informed consent)
* Affiliate or beneficiary of a social security scheme

Exclusion Criteria:

* Patients with non-idiopathic carpal tunnel syndrome with medical contraindication : pregnancy, obesity (body mass index > 30), diabetes, rheumatoid arthritis, sarcoidosis, purulent tenosynovitis, tuberculosis, systemic lupus erythematosus, hypothyroidism or hyperthyroidism and gout.
* Patients with history of cardiac disease or coronary artery disease.
* Patients with systemic amyloidosis already known.
* Patients unde guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Interventional transversal monocentric study with prospective recruitment.
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
Cardiac involvement | 1 day
  Prevalence of cardiac involvement in presence of transthyretin amyloid deposition in the transverse carpal ligament of patients with CTS referred for surgery released.

SECONDARY OUTCOMES:
Transthyretin amyloid involvement | 1 day
  Prevalence of transthyretin amyloid deposition in the transverse carpal ligament of patients with CTS referred for surgery released. Electrocardiographic features of cardiac involvement in case of presence of transthyretin amyloid deposition in the transverse carpal ligament of patients with CTS referred for surgery released.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier LAIREZ, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Olivier Lairez, Toulouse, France